CLINICAL TRIAL: NCT02726568
Title: A Phase II Study to Determine the Efficacy and Safety of High Dose Icotinib Combined With Stereotatic Radiosurgery for NSCLC Patients Harboring EGFR Mutation With Brain Metastases
Brief Title: High Dose Icotinib With Sequential SRS For NSCLC Patients Harboring EGFR Mutation With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV-65
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Non-small Cell Lung Cancer; Brain Metastases
Keywords: EGFR-TKI; NSCLC; Icotinib; SRS; radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Icotinib 375mg Tid (Experimental): The human subject gets icotinib 375mg, Tid until intracranial PD or intolerable toxicity reaction.
  Interventions: Drug: Icotinib; Radiation: SRS

INTERVENTIONS:
Drug: Icotinib — 375 mg Tid (1125 mg per day) until intracranial PD.
Radiation: SRS — If intracranial PD, then the subjects get stereotatic radiosurgery （30Gy/3f) combined with Icotinib 375mg Tid.

SUMMARY:
This trail is designed to assess the efficacy and safety of high dose Iconitib combined with SRS for NSCLC patients harboring EGFR mutation with brain metastases.

DETAILED DESCRIPTION:
The long-term control of brain metastases becomes a clinical challenge. Whole brain radiotherapy, the standard treatment for patients with multiple brain metastases, can only bring a modest survival improvement around 3-6 months. EGFR-TKIs like icotinib with its proven activity in non-small cell lung cancer may provide clinical benefits to brain metastases patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of non-small cell lung cancer (NSCLC);
* Diagnosis of brain metastases on a Gadolinium-enhanced MRI.
* Less than 10 sites of intracranial metastases, or the longest diameter of the intracranial lesion is less than 4cm.
* Positive EGFR mutation（Ex19del or 21L858R）.
* Life expectancy ≥3months.
* Have one or more measurable encephalic lesions according to RECIST.
* The patient has not received radiotherapy for the head or extracranial target lesions before.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L.
* Adequate renal function: Serum creatinine ≤1.5 x ULN, or ≥ 50 ml/min.
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) and Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases.
* Female subjects should not be pregnant.
* All human subjects should able to comply with the required protocol and follow-up procedures, and able to receive oral medications.
* Written informed consent provided.

Exclusion Criteria:

* Previous usage of EGFR-TKI or antibody to EGFR: gefitinib, erlotinib, herceptin, erbitux.
* CSF or MRI findings consistent with metastases of spinal cord, meninges or meningeal.
* Allergic to Icotinib.
* Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active peptic ulcer disease.
* Pregnancy or breast-feeding women.
* Participate in the other anti-tumor clinical trials in 4 weeks.
* have quit from the trail before.
* Any other serious underlying medical, psychological and other condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
intracranial progression-free survival | from date of randomization until the date of first documented intracranial progression, assessed up to 12 months.

SECONDARY OUTCOMES:
progress-free survival | from date of randomization until the date of extracranial progression, assessed up to 18 months.
overall survival | from date of randomization until the date of death, assessed up to 36 months.
objective response rate | from date of randomization until the date of progression, assessed up to 12 months.
disease control rate | from date of randomization until the date of progression, assessed up to 18 months.
Quality of life measured by FACT-L/LCS 4.0 and FACT-Br | from date of randomization until the date of death from any cause, assessed up to 36 months.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by NCI-CJ-CAE3.0 | from date of randomization until the date of death, assessed up to 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: YOU LU, M.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided